CLINICAL TRIAL: NCT04461691
Title: Cryoballoon Pulmonary Vein Isolation for Atrial Fibrillation With Heart Failure
Acronym: POLAR-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Josefs-Hospital Wiesbaden GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLAR-HF
Record Dates: First submitted 2020-05-08; First posted 2020-07-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Heart Failure; Cryoballon Ablation
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart Failure (Other): Cryoballoon pulmonary vein isolation is a common method for catheter ablation of atrial fibrillation. Cryoenergy is applied through a balloon in a single-step approach resulting in necrosis by tissue freezing.
  Interventions: Procedure: Cryoballoon Pulmonary Vein Isolation
- Normal cardiac function (Other): Cryoballoon pulmonary vein isolation is a common method for catheter ablation of atrial fibrillation. Cryoenergy is applied through a balloon in a single-step approach resulting in necrosis by tissue freezing.
  Interventions: Procedure: Cryoballoon Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Cryoballoon Pulmonary Vein Isolation — Cryoballoon pulmonary vein isolation is a common method for catheter ablation of atrial fibrillation. Cryoenergy is applied through a balloon in a single-step approach resulting in necrosis by tissue freezing.

SUMMARY:
The combination of atrial fibrillation (AF) and heart failure (HF) is common and implies a poor prognosis. Pulmonary vein isolation is an established method for the treatment of symptomatic AF in patients with normal heart function and has been shown to be more effective than drug therapy. Recently, radiofrequency ablation has shown a positive effect in patients with AF and HF. POLAR-HF has been designed to investigate efficacy and safety of cryoballoon pulmonary vein isolation in patients with paroxysmal or persistent AF and severe HF (LVEF ≤ 40%).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal or persistent atrial fibrillation
* Patients with severe heart failure (LVEF ≤40%, assigned to heart failure group)
* Patients with normal cardiac function (assigned to control group)
* Age > 18 years
* Consent capacity

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Lack of consent capacity

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1420 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures (Number of recurrence) | 60 months
  Number of subjects with recurrence of atrial fibrillation, atrial flutter, atrial tachycardia or re-ablation after a blanking Period of 90 days after the initial cryoablation procedure
Primary Outcome Measures (number of safety events) | 60 months
  2. Number of subjects with a primary safety event including a composite of death from any cause, stroke or transient ischemic attack and serious procedure-related adverse events (Major Bleeding by International Society on Thrombosis and Hemostasis (ISTH) criteria, pericardial effusion, cerebrovascular or systemic embolism, phrenic paresis, major groin site complications requiring treatment)

SECONDARY OUTCOMES:
Secondary Outcome Measures (number of deaths) | 60 months
  Number of all-cause death
Secondary Outcome Measures (procedural success) | 60 months
  2. Incidence of acute procedural success assessed by successful isolation of all pulmonary veins
Secondary Outcome Measures (rehospitalization) | 60 months
  3. Number of subjects reporting a first unplanned rehospitalization for cardiovasvular causes
Secondary Outcome Measures (procedure duration) | 60 months
  4. Total procedure duration and left-atrial dwell time (in minutes)
Secondary Outcome Measures (total time) | 60 months
  5. Total fluoroscopy time (in minutes)
Secondary Outcome Measures (total contrast use) | 60 months
  6. Total contrast dye use (in milliliters)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Ehrlich, MD, Principal Investigator — St. Josefs-Hospital Wiesbaden GmbH; Andreas Boehmer, MD, Principal Investigator — St. Josefs-Hospital Wiesbaden GmbH
Locations (1):
- St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden, Germany

REFERENCES:
- [Derived] Boehmer AA, Rothe M, Andrade JG, Wiedenmann L, Spork P, Schneider KY, Nussbaum E, Keim C, Weiss P, Dobre BC, Feickert S, Ruckes C, Dyrda K, Kaess BM, Nattel S, Ehrlich JR. Pulmonary Vein Isolation Only for Atrial Fibrillation With Heart Failure (POLAR-HF). JACC Clin Electrophysiol. 2025 Nov 19:S2405-500X(25)00812-6. doi: 10.1016/j.jacep.2025.09.041. Online ahead of print. PMID 41263723